CLINICAL TRIAL: NCT00597480
Title: Study of Growth-promoting and Metabolic Effects of Growth Hormone (rhGH) by Comparison of Two Regimens of rhGH Administration to SGA Children. Pharmacogenetics of Metabolic Responses to rhGH
Brief Title: Study of Growth-promoting and Metabolic Effects of Growth Hormone (rhGH)
Acronym: SGA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no more inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070303
Record Dates: First submitted 2008-01-07; First posted 2008-01-18 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Small for Gestational Age
Keywords: Growth hormone; Child; insulin resistance; metabolic syndrome X; children born small for gestational age
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): the recommended dose in the EU of rhGH (Norditropine SimpleXx®)
  Interventions: Drug: rhGH (Norditropine SimpleXx®)
- 2 (Active Comparator): the dose to achieve a "treat-to target" value of IGF-1 levels within a +1.5 to +2.5 SDS interval (starting dose, 0.067 mg/kg/day)
  Interventions: Drug: rhGH norditropine simple Xx

INTERVENTIONS:
Drug: rhGH (Norditropine SimpleXx®) — the recommended dose in the EU of rhGH (Norditropine SimpleXx®
  Arms: 1
Drug: rhGH norditropine simple Xx — the dose to achieve a "treat-to target" value of IGF-1 levels within a +1.5 to +2.5 SDS interval (starting dose, 0.067 mg/kg/day)
  Arms: 2

SUMMARY:
Recombinant growth hormone (rhGH) treatment is widely used in France to normalize height during childhood and final height in children born small for gestational age (SGA). Because rhGH has been associated with increased insulin levels and insulin resistance, concern has been expressed regarding the late consequences of rhGH treatment on risk factors for diabetes mellitus type II and metabolic syndrome, especially in possibly predisposed subjects as SGA children.

DETAILED DESCRIPTION:
Recombinant growth hormone (rhGH) treatment is widely used in France to normalize height during childhood and final height in children born small for gestational age (SGA). Because rhGH has been associated with increased insulin levels and insulin resistance, concern has been expressed regarding the late consequences of rhGH treatment on risk factors for diabetes mellitus type II and metabolic syndrome, especially in possibly predisposed subjects as SGA children.

Because rhGH use in this population will sharply increase in the coming years, our purpose is to identify and analyze factors that predispose these children born SGA to the metabolic consequences of rhGH therapy.

The main objective of this study is to identify and analyze factors implicated in the variability of the metabolic and growth responses to rhGH treatment in children born SGA. We want to:

* Quantify the metabolic effects of rhGH treatment by analyzing insulin levels, insulin sensitivity and lipid profile (lipolysis and ketogenesis);
* Evaluate the effects of two different rhGH regimens on the growth of children born SGA;
* Determine if the metabolic effects of rhGH therapy correlate to the growth responses in the two groups;
* Identify factors, especially genetic factors, responsible for the variations in individual metabolic and growth-promoting effects of rhGH in children born SGA.

This is a randomized, open-labeled, 2-year study, which will compare two regimens of rhGH therapy on the growth responses and metabolic effects in short children born SGA.

100 prepubertal, non GH deficient, short children (height < -3 SDS) born SGA (birth height < -2 SDS) will be randomized to receive either the recommended dose in the EU of rhGH (Norditropine SimpleXx®), or the dose to achieve a "treat-to target" value of IGF-1 levels within a +1.5 to +2.5 SDS interval (starting dose, 0.067 mg/kg/day) for 24 months.

Metabolic effects of rhGH treatment will be evaluated by body mass index (BMI), fasting insulin and glucose levels, HOMA index of insulin resistance, insulin and glucose levels during OGTT, HbA1C and fasting serum lipids (free fatty acids, 3-hydroxybutyrate, total cholesterol, LDL and HDL cholesterol, triglycerides). Height, growth velocity, IGF-1 and IGF-BP3 levels will evaluate growth response of rhGH treatment.

Polymorphisms of different genes of the signaling pathway of GH and insulin will be analyzed in order to search for those possibly responsible for the variability in metabolic and growth responses during rhGH treatment in SGA children.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal age
* Prepubertal characteristics
* Non GH deficient
* Short children (height < -2.5 SDS)
* Born SGA (birth height < -2 SDS)
* Parental height adjusted (< -1 DS)
* No rhGH treatment before inclusion

Exclusion Criteria:

* ALLERY to rhGH or excipients
* Small height etiologies
* Cancer or cancer treatment ongoing
* Drugs interference with growth
* Mental impairment
* Hypertrophic cardiopathy impairment
* Hypertension not under controlled
* Intra cranial hypertension not controlled
* Diabetes and hyperglycaemia without diabetes
* Dyslipidemia
* Hepatitis
* Kidney failure
* Chromosomic aberration and/or genetic disorders (except Silver Russel Syndrome)
* No social security
* State of health in worst conditions after cardiac surgery, polytraumatism

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Identify and analyze factors implicated in the variability of the metabolic and growth responses to rhGH treatment in children born SGA | every three months during twenty seven months

SECONDARY OUTCOMES:
Metabolic effects of rhGH treatment will be evaluated by body mass index (BMI) | every three months during
Polymorphisms of different genes of the signaling pathway of GH and insulin | the day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Teinturier, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Saint Vincent de Paul, Paris, France